CLINICAL TRIAL: NCT04214639
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Vehicle Controlled, Parallel-Group, Clinical Study Comparing the Efficacy and Safety of IDP-126 Gel in the Treatment of Acne Vulgaris
Brief Title: Clinical Study Comparing the Efficacy and Safety of IDP-126 Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V01-126A-301
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDP-126 Gel (Experimental)
  Interventions: Drug: IDP-126 Gel
- IDP-126 Vehicle Gel (Placebo Comparator)
  Interventions: Drug: IDP-126 Vehicle Gel

INTERVENTIONS:
Drug: IDP-126 Gel — IDP-126 Gel applied topically to the face once daily for 12 weeks.
  Arms: IDP-126 Gel
Drug: IDP-126 Vehicle Gel — IDP-126 Vehicle Gel applied topically to the face once daily for 12 weeks.
  Arms: IDP-126 Vehicle Gel

SUMMARY:
This is a multicenter, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, tolerability, and efficacy of IDP-126 Gel in comparison IDP-126 Vehicle Gel at Weeks 2, 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 9 years of age and older.
* Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit).
* Subject must have an Evaluator's Global Severity Score (EGSS) of 3 (moderate) or 4 (severe) at the baseline visit.
* Subjects with a facial acne inflammatory lesion (papules, pustules, and nodules) count no less than 30, but no more than 100.
* Subjects with a facial acne non-inflammatory lesion (open and closed comedones) count no less than 35, but no more than 150.
* Subjects with 2 or fewer facial nodules.

Exclusion Criteria:

* Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram negative folliculitis, dermatitis, eczema.
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
* Subjects with more than 2 facial nodules.
* Female subjects who are pregnant, nursing mothers, planning a pregnancy during the course of the study, or become pregnant during the study.
* Use of estrogens (eg, Depogen, Depo-Testadiol, Gynogen, Valergen, etc) for less than 12 weeks immediately preceding study entry; subjects treated with estrogens 12 or more consecutive weeks immediately prior to study entry need not be excluded unless the subject expects to change dose, drug or discontinue estrogen use during the study.
* Treatment of any type of cancer within the last 6 months, with the exception of complete surgical excision of skin cancer outside the treatment area.
* Subjects who have not undergone specified washout period(s) for topical preparations/physical treatments used on the face or subjects who require the concurrent use in the treatment area.
* Subjects who have not undergone specified washout period(s) for systemic medications or subjects who require the concurrent use of systemic medications.
* Subjects with any underlying disease that the investigator deems uncontrolled, and poses a concern for the subject's safety while participating in the study.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health
Locations (13):
- United States (11):
  - Bausch Site 110, Bryant, Arkansas
  - Bausch Site 104, Fremont, California
  - Bausch Site 109, Denver, Colorado
  - Bausch Site 102, Boynton Beach, Florida
  - Bausch Site 111, North Miami Beach, Florida
  - Bausch Site 106, Sanford, Florida
  - Bausch Site 103, Las Vegas, Nevada
  - Bausch Site 114, New York, New York
  - Bausch Site 105, High Point, North Carolina
  - Bausch Site 107, Nashville, Tennessee
  - Bausch Site 108, Pflugerville, Texas
- Canada (2):
  - Bausch Site 101, Barrie, Ontario
  - Bausch Site 113, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gold M, Lain T, Harper JC, Baldwin H, Guenin E, Stein Gold L. Efficacy and Safety of Clindamycin Phosphate 1.2%/Adapalene 0.15%/Benzoyl Peroxide 3.1% Gel: Post Hoc Analysis by Baseline Disease Severity. Dermatol Ther (Heidelb). 2025 Jul;15(7):1867-1882. doi: 10.1007/s13555-025-01440-z. Epub 2025 May 16. PMID 40377868
- [Derived] Kircik LH, Stein Gold L, Gold M, Weiss JS, Harper JC, Del Rosso JQ, Bunick CG, Bhatia N, Tanghetti EA, Eichenfield LF, Baldwin H, Draelos ZD, Callender VD, Han G, Gooderham MJ, Sadick N, Lupo MP, Lain ET, Werschler WP. Triple Combination Clindamycin Phosphate 1.2%/Adapalene 0.15%/Benzoyl Peroxide 3.1% for Acne: Efficacy and Safety from a Pooled Phase 3 Analysis. Dermatol Ther (Heidelb). 2024 May;14(5):1211-1227. doi: 10.1007/s13555-024-01155-7. Epub 2024 May 9. PMID 38724841

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel
Started | 122 | 61
Completed | 107 | 55
Not Completed | 15 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel | Total
Number analyzed (Participants) | 122 | 61 | 183
Age, Continuous [Median (Full Range); unit: years] | 17 [10 to 42] | 18 [12 to 44] | 17 [10 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 31 | 106
  Male | 47 | 30 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 4 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 28 | 9 | 37
  White | 75 | 45 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Baseline Evaluator's Global Severity Score [Count of Participants; unit: Participants] — The Evaluator's Global Severity Score has grades for acne severity of 0 (Clear), 1 (Almost Clear), 2 (Mild), 3 (Moderate), and 4 (Severe), with higher scores indicating worse severity.
  Participants
    Moderate | 107 | 58 | 165
    Severe | 15 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline to Week 12 in Inflammatory Lesion Counts
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Deviation); unit: lesion counts
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel
Number analyzed (Participants) | 122 | 61
lesion counts | -27.7 (9.55) | -21.7 (8.79)

2. Primary Outcome: Absolute Change From Baseline to Week 12 in Non-inflammatory Lesion Counts
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Deviation); unit: lesion counts
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel
Number analyzed (Participants) | 122 | 61
lesion counts | -35.4 (15.52) | -23.5 (14.93)

3. Primary Outcome: Percentage of Participants With Success on the Evaluator's Global Severity Score
Description: Success was defined as at least a two grade reduction and clear or almost clear at Week 12. The Evaluator's Global Severity Score has grades for acne severity of 0 (Clear), 1 (Almost Clear), 2 (Mild), 3 (Moderate), and 4 (Severe), with higher scores indicating worse severity.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel
Number analyzed (Participants) | 122 | 61
percentage of participants | 49.6 | 24.9

4. Secondary Outcome: Inflammatory Lesion Count Percentage Changes at Week 4, 8, and 12
Time Frame: Baseline to Week 4, 8, 12
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel
Number analyzed (Participants) | 122 | 61
percentage change
  Week 4 | -51.14 (26.115) | -38.91 (25.691)
  Week 8 | -63.35 (27.793) | -50.58 (26.569)
  Week 12 | -75.70 (26.663) | -59.62 (24.348)

5. Secondary Outcome: Noninflammatory Lesion Count Percentage Changes at Week 4, 8, and 12
Time Frame: Baseline to Week 4, 8, 12
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel
Number analyzed (Participants) | 122 | 61
percentage change
  Week 4 | -45.87 (28.119) | -30.42 (27.455)
  Week 8 | -57.92 (31.654) | -44.70 (30.118)
  Week 12 | -72.70 (32.364) | -47.61 (31.069)

6. Secondary Outcome: Percentage of Participants With at Least a Two Grade Reduction on the Evaluator's Global Severity Score at Week 12
Description: The Evaluator's Global Severity Score has grades for acne severity of 0 (Clear), 1 (Almost Clear), 2 (Mild), 3 (Moderate), and 4 (Severe), with higher scores indicating worse severity.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel
Number analyzed (Participants) | 122 | 61
percentage of participants | 57.2 | 24.8

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/61
Other Adverse Events (participants affected / at risk) | 17/122 | 0/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-126 Gel (N=122) | IDP-126 Vehicle Gel (N=61)
Application site pain (General disorders) | 15 | 0
Erythema (Skin and subcutaneous tissue disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT04214639/Prot_SAP_000.pdf